CLINICAL TRIAL: NCT03782753
Title: Longitudinal Study of Molecular Pathology and Neuronal Networks in Leucine-rich Repeat Kinase 2 Carriers and Idiopathic Parkinson's Disease Patients and Healthy Controls Using PET, MR Imaging, and Other Markers of in Vivo Pathology
Brief Title: Molecular Pathology and Neuronal Networks in LRRK2 Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 249061
Record Dates: First submitted 2018-12-14; First posted 2018-12-20 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease, PARK8; Parkinson Disease; Idiopathic Parkinson Disease
Keywords: Parkinson Disease; LRRK2
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 8

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: 25 LRRK2-PD patients
- Group B: 25 idiopathic PD patients
- Group C: 25 HC subjects

SUMMARY:
Parkinson's Disease (PD) is a progressive neurodegenerative disease characterized clinically by bradykinesia, resting tremor, rigidity, and postural instability. Little is known about the mechanisms underlying neuronal degeneration in PD and currently, no treatment is available to halt disease progression in PD.

The pathophysiological characterisation of phenomena occurring in the time window between the pathological start of the disease and the onset of motor symptoms is crucial to develop potential neuroprotective agents.

Several genes have been discovered providing important insights on the pathogenesis of PD. Mutations of Leucine-rich repeat kinase 2 (LRRK2) are associated with 2-5% of all PD cases in North American Caucasians. LRRK2 is an enzyme that in humans is encoded by the autosomal dominant Parkinson's disease-8 (PARK8) gene, which is associated with an increased risk of PD.

Clinical and digital biomarkers, blood and cerebrospinal fluid (CSF) biomarkers and molecular positron emission tomography (PET) imaging, with specific radioligands, provide invaluable insights to help understand and characterise disease pathophysiology.

The investigators aim to characterize molecular phenomena underlying LRRK2 PD with the hope of providing further insights into possible mechanisms taking place in PD and to help identify targets for disease-modifying therapeutics.

ELIGIBILITY:
Inclusion Criteria:

All groups

* Women of child-bearing potential must use protocol-defined contraceptive measures and must have a negative β-hCG test at screening. For sexually active subjects (except females of non-childbearing potential), condoms should be used in addition to other birth control methods during the study, for 15 days after the last dose of investigational drug, and for 3 months after the last administration of PET or SPECT ligands. All male subjects must agree to refrain from donating sperm during the study, for 15 days following the last dose of investigational drug, and for 3 months after the last administration of PET or SPECT ligands. It is important that male subjects not impregnate others while in the study.
* Adequate visual and auditory acuity to complete the psychological testing.

Idiopathic PD group

* Clinical diagnosis of Parkinson's disease meeting the Movement Disorder Society Clinical Diagnostic Criteria (i.e. not induced by drugs or other diseases or carriers of PD risk genes such as LRRK2, SNCA, PARK2 etc.).
* Hoehn and Yahr scale stage 1 or 2.
* Patients who are drug-naïve (never been treated with dopamine agonists or levodopa) or on dopamine replacement therapy.
* Patients who have received the diagnosis of idiopathic PD within three years for drug-naïve patients or within eight years for patients on dopamine replacement therapy.

LRRK2 PD group

* Clinical diagnosis of Parkinson's disease meeting the Movement Disorder Society Clinical Diagnostic Criteria and genetic confirmation of being carriers of LRRK2 PD risk genes, diagnosed after the age of 30 years.
* Hoehn and Yahr scale stage 1 or 2.
* Patients who are drug-naïve (never been treated with dopamine agonists or levodopa) or on dopamine replacement therapy.
* Patients who have received the diagnosis of idiopathic PD within three years for drug-naïve patients or within eight years for patients on dopamine replacement therapy.

Exclusion Criteria:

* Patients who had previous surgery for PD (including but not limited to deep brain stimulation [DBS] or cell transplantation).
* Patients who are treated with duodopa or apomorphine.
* Patients taking serotonin acting drugs such as antidepressants (i.e. tricyclic or selective serotonin reuptake inhibitors etc.)
* Patients taking drugs acting on SV2A such as antiepileptics (i.e. levetiracetam or brivaracetam etc.)
* Pregnancy or breastfeeding.
* Patients with current or a recent history of drug or alcohol abuse/dependence.
* Patients who have other neurological disorders and known intracranial co-morbidities such as stroke, haemorrhage, space-occupying lesions.
* Presence of any clinically significant medical condition (including cardiovascular, respiratory, cerebrovascular, hematological, hepatic, renal, gastrointestinal, or other disease) that, based on the judgment of the investigator, is clinically unstable, is likely to deteriorate during the course of the study, could put the patient at risk because of participation in the study, could affect the subject's ability to complete the study, or could influence the study results.
* History of suicidal behavior or active suicidal ideation.
* Within 1 year prior to screen or between screen and baseline (Day -1), any of the following: myocardial infarction; hospitalization for congestive heart failure; hospitalization for, or symptoms of, unstable angina; or syncope not related to PD.
* History or presence of renal disease or impaired renal function.
* Clinically important infection (e.g., chronic, persistent, or acute infection) within 30 days prior to screen or between screen and baseline (Day -1).
* History of cancer within the last 5 years, with the exception of nonmetastatic basal cell carcinoma of the skin.
* Clinically significant blood clotting or bleeding disorder, including clinically significant abnormal findings in laboratory assessments of coagulation or hematology.
* Use of antipsychotic medication within 3 months prior to screen or between screen and baseline (Day -1).
* Use of any anticoagulant within 30 days prior to baseline PET scan.
* Use of any oral corticosteroid within 30 days prior to baseline PET scan.
* Use of metoclopramide within 30 days prior to baseline (Day -1).
* Use of any thyroid medication within 30 days prior to baseline (Day -1).
* Regular use (e.g., taken > 3 days/week) of narcotic pain medications within 30 days prior to baseline (Day -1).
* Presence of any of the following MRI contraindications: pacemaker; cardiac defibrillator; spinal cord or vagus nerve stimulator; aneurysm clip; artificial heart valve; recent coronary or carotid stent; ear implant; CSF shunt; other implanted medical device (e.g., Swan-Ganz catheter, insulin pump); or metal fragments or foreign objects in the eyes, skin, or body.
* Negative Allen test in both hands, unless the brachial artery is used for arterial cannulation.
* Claustrophobia and history of back pain that makes prolonged laying on the PET or MRI scanner intolerable.
* Initiation or change in pharmacologic therapy for symptoms of PD within 30 days prior to screen or between screen and baseline (Day -1).

In addition, the following are exclusionary for subjects participating in CSF sampling:

- Any spinal malformations or other aspects (e.g., tattoos) or other clinical findings (e.g., papilledema seen with ophthalmoscopy) that may complicate or contraindicate lumbar puncture, as judged by the investigator.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: LRRK2 PD patients, idiopathic PD patients and healthy controls.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Changes in serotonergic transmission in the ventral and dorsal raphe nuclei, and in raphe projection areas, in LRRK2-PD compared to idiopathic PD. | One year
  The study's main outcome measure is changes in serotonergic neurotransmission within specific brain regions. This will be assessed with positron emission tomography (PET) imaging using the readioligand 11C-labeled 3-amino-4 -(2-dimethylaminomethyl-phenylsulfanyl)benzonitrile ([11C]DASB).

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom